CLINICAL TRIAL: NCT07386834
Title: The Effect of Oro-esophageal Versus Nasogastric Feeding for Stroke Patients With Dysphagia: A Multicenter Randomized Controlled Large-Scale Study
Brief Title: Large-Scale Study of Oro-esophageal Feeding Versus Nasogastric Feeding for Swallowing Function and Airway Protection
Acronym: IOEfinal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Principle Investigator, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IOElastreport
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oro-esophageal Group (Experimental): Participants will receive oro-esophageal feeding plus rehabilitation therapy in accordance with stroke rehabilitation guidelines, with the specific content determined by the participating centers, for 14 days and being hospitalized.
  Interventions: Dietary Supplement: Oro-esophageal Feeding; Behavioral: Rehabilitation care
- Nasogastric Group (Active Comparator): Participants will receive Nasogastric feeding plus rehabilitation therapy in accordance with stroke rehabilitation guidelines, with the specific content determined by the participating centers, for 14 days and being hospitalized.
  Interventions: Dietary Supplement: Nasogastric Feeding; Behavioral: Rehabilitation care

INTERVENTIONS:
Dietary Supplement: Oro-esophageal Feeding — Medical staff inserts the tube slowly and smoothly into the upper esophagus, verifying the correct insertion depth by referencing the calibration marks on the tube wall. The distance from the incisors to the tube's tip should range from 22 to 25 cm. Following insertion, the distal end of the tube is submerged in a container of water, and the absence of continuous bubbling confirms successful intubation. Feeding is subsequently administered three times daily at a rate of 50 mL per minute, with a volume of 400 to 600 mL per feeding. The intervention period lasts for a total of two weeks.
  Arms: Oro-esophageal Group
Dietary Supplement: Nasogastric Feeding — The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups.The intervention period lasts for a total of two weeks.
  Arms: Nasogastric Group
Behavioral: Rehabilitation care — All patients will receive rehabilitation care according to the standard of care for the trial site hospital. All these interventions are performed in accordance with the Chinese Guidelines for Stroke Rehabilitation and the Chinese Guidelines for Dysphagia Rehabilitation. The intervention period lasts for a total of two weeks.

SUMMARY:
This is a randomized controlled trial involving patients with ischemic stroke and dysphagia. The aim of this study is to explore the recovery speed and therapeutic effect of oro-esophageal feeding compared with nasogastric feeding on swallowing function. This study mainly addresses the following two research questions: 1. Whether oro-esophageal feeding improves swallowing function more rapidly and effectively than nasogastric tube feeding. 2. Whether oro-esophageal feeding is non-inferior to nasogastric tube feeding in terms of safety.

DETAILED DESCRIPTION:
This is a randomized controlled trial involving patients with ischemic stroke and dysphagia. The aim of this study is to explore the recovery speed and therapeutic effect of oro-esophageal feeding compared with nasogastric feeding on swallowing function. This study mainly addresses the following two research questions: 1. Whether oro-esophageal feeding improves swallowing function more rapidly and effectively than nasogastric tube feeding. 2. Whether oro-esophageal feeding is non-inferior to nasogastric tube feeding in terms of safety.

The intervention period will last for two weeks, with an additional four-week follow-up observation period. This is a multicenter study to be conducted across multiple hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* First stroke
* Disease duration less than one month.
* Ischemic stroke.
* Patients who need enteral feeding.
* Dysphagia confirmed by imaging Study.
* Clear consciousness.
* Stable vital signs.
* With informed consent and participants who understand and agree to comply with planned study procedures.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases or structural abnormalities.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Contraindications for tube feeding.
* Pregnancy or breast feeding.
* Anticipated discharge from the hospital or transfer to another hospital within one week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale | Day 0 and day15
  The Dysphagia Outcome and Severity Scale consists of 7 levels, from 1 to 7, based on imaging data. A higher level indicates better swallowing function.

SECONDARY OUTCOMES:
Time to improvement of one level and of the baseline Dysphagia Outcome and Severity Scale | up to 2 weeks
  The Dysphagia Outcome and Severity Scale consists of 7 levels, from 1 to 7, based on imaging data.
  The investigators will record the time required for participants to achieve a one-grade improvement from the baseline Dysphagia Outcome and Severity Scale.
Time to oral intake | up to 2 weeks
  The time to recovery is the first day, during the two weeks of the intervention period, on which a participant meets level 3, 4, 5, 6, or 7 on the Dysphagia Outcome and Severity Scale. The Dysphagia Outcome and Severity Scale consists of 7 levels, from 1 to 7, based on imaging data. A higher level indicates better swallowing function.
Penetration-Aspiration Scale | Day 0 and day15
  The Penetration-Aspiration Scale is for assessing airway protection. It has 8 grades, grouped into 3 categories: no penetration/aspiration, penetration, aspiration. Lower grades = better function: Grade 1 is optimal (no airway entry); Grade 8 is most severe (food enters airway below vocal cords with no clearing effort).
Murray Secretion Scale | Day 0 and day15
  The Murray Secretion Scale is used to evaluate the accumulation of secretions, in which grade 0 meant no obvious accumulation, and grade 3 meant secretions in the laryngeal vestibule. The Murray Secretion Scale has 4 grades. The higher grade indicates more severe accumulation of secretions.
Yale Pharyngeal Residual Severity Rating Scale | Day 0 and day15
  The Yale Pharyngeal Residual Severity Rating Scale is used to evaluate pharyngeal residue after swallowing. The score could range between 1 and 5, with higher scores indicating worse situations.
Aspiration | up to 6 weeks
  Aspiration is based on self-reporting, caregiver monitoring, or the diagnosis of aspiration pneumonia, defined as the coughing and discomfort caused by food or water entering the airway for various reasons. The numbers of aspiration will be recorded.